CLINICAL TRIAL: NCT01701193
Title: A Randomized Double-Blind Controlled Proof-of-Concept Study of Alanyl-Glutamine for Reduction of Post-Myomectomy Adhesions
Brief Title: A Clinical Study of Alanyl-Glutamine for Reduction of Post-Myomectomy Adhesions
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Temple Therapeutics BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Ade002; NCT04250467 (obsolete NCT alias)
Record Dates: First submitted 2012-10-03; First posted 2012-10-05 (Estimated); Results first posted 2021-05-07 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-03

CONDITIONS: Pelvic Adhesions
MeSH Terms: interventions — alanylglutamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Physiological saline- Laparoscopic (Placebo Comparator): Participants receiving intraperitoneal administration of physiological saline at the time of laparoscopic myomectomy.
  Interventions: Drug: Physiologic saline
- L-Alanyl/L-Glutamine- Laparoscopic (Experimental): Participants receiving intraperitoneal administration of L-Alanyl-L-Glutamine at the time of laparoscopic myomectomy.
  Interventions: Drug: L-Alanyl/L-Glutamine
- Physiological saline- Laparotomy (Placebo Comparator): Participants receiving intraperitoneal administration of physiological saline at the time of myomectomy (laparotomy).
  Interventions: Drug: Physiologic saline
- L-Alanyl/L-Glutamine- Laparotomy (Experimental): Participants receiving intraperitoneal administration of L-Alanyl-L-Glutamine at the time of myomectomy (laparotomy).
  Interventions: Drug: L-Alanyl/L-Glutamine

INTERVENTIONS:
Drug: L-Alanyl/L-Glutamine — Sterile solution of L-Alanyl-L-Glutamine, 400mg/mL in water for injection. It is dosed at 1g/kg of body weight and is instilled into the peritoneum at the time of surgery. The active ingredient, glutamine, is a conditionally essential amino acid component of nutritional supplements.
  Other Names: Evitar
  Arms: L-Alanyl/L-Glutamine- Laparoscopic; L-Alanyl/L-Glutamine- Laparotomy
Drug: Physiologic saline — Placebo
  Arms: Physiological saline- Laparoscopic; Physiological saline- Laparotomy

SUMMARY:
This study evaluates whether L-Alanyl-L-Glutamine can reduce the incidence, extent and severity of adhesions after myomectomy. Half of the participants will receive L-Alanyl-L-Glutamine and the other half of participants will receive a saline placebo at the time of myomectomy.

DETAILED DESCRIPTION:
The myriad medical and financial burdens of post-operative adhesions are well documented; however, treatment options are limited and controversial. Implantable physical barriers to prevent adhesions are commercially available, but most trials have failed to demonstrate compelling evidence to support widespread use. In recent years, advances have been made in our understanding of the cellular mechanisms underlying adhesiogenesis, raising the prospect of targeting these pathways to prevent post-surgical adhesions. However, to date, no drug has received regulatory approval for this purpose in any jurisdiction. Our study was designed to evaluate the efficacy and safety of a single intraoperative intraperitoneal dose of L-Alanyl-L-Glutamine (AG), an agent which has been shown to act upon key mediators in the adhesion formation pathway.

Methods: This was a randomized, double-blind, placebo-controlled study (DBRCT) of 47 women who underwent myomectomies by laparoscopy (N=37; AG-18 vs Placebo-19) or laparotomy (N=10; AG-5 vs Placebo-5) with a scheduled clinically necessary second-look laparoscopy (SLL) 6 - 8 weeks later. Digital recordings were obtained for all procedures. The primary endpoint was reduction in the incidence, severity and extent of post-operative adhesions, as analyzed by intention-to-treat (ITT) approach.

Three independent, blinded reviewers evaluated the operative video recordings to assess for presence of adhesions. Secondary endpoints assessed the safety and tolerability of AG. Post-hoc analysis assessed presence or absence of adhesions in the peritoneal cavity. Patients included those with previous history of surgery, endometriosis, and adhesiolysis was permitted at myomectomy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are female
* Subjects are 18 years of age or older at the time of consent
* Subjects have a BMI between 17-40
* Subjects must have signed informed consent form
* Subjects have a preoperative diagnosis of uterine fibroids and plan to have a myomectomy completed surgically as part of their standard of care
* Subjects must have a physical examination and compliance assessment

Exclusion Criteria:

* Subjects whose BMI is outside the range of 17-40
* Subjects participating in another clinical trial with a drug or device
* Subjects who have participated in a clinical trial with a drug or device within 30 days prior to this study
* Subjects with suspected or diagnosed pregnancy
* Subjects with suspected intraabdominal infection
* Subjects who are immunocompromised
* Subjects diagnosed with cancer
* Subjects treated with hemostatic agents (e.g. fibrin sealant, collagen, oxidized cellulose)
* Subjects treated with adhesion prevention agents other than the Anti-Adhesion product (APP) (e.g. Intergel ® Adhesion Prevention Solution, Seprafilm ® Membrane)
* Subjects taking anti-epileptic medication
* Subjects who have been treated with Methotrexate or other chemotherapeutics agents
* Subjects with an American Fertility Society score of Stage D at the time of myomectomy as determined by the surgeon
* Positive viral serology screening results for hepatitis B surface antigen, antibodies to hepatitis C virus or human immunodeficiency

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2015-02-15 (Actual); Primary Completion 2016-10-20 (Actual); Study Completion 2016-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donna Chizen, MD, FRCSC, Principal Investigator — University of Saskatchewan
Locations (1):
- 8Surgery and Endoscopy Department of Kharkiv Medical Academy of Postgraduate Education Kharkiv City Clinical Multi-field Hospital, Kharkiv, Ukraine

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a single-center study at a private hospital clinic. Recruitment was between February 2015 and October 2016. Subjects were adult women planned for myomectomy with a scheduled clinically necessary second look laparoscopy. The study and consent form were approved by the Institutional Review Board/Ethics Committee and the Investigator's IRB/EC (Ethics Committee of Kharkiv City Clinical Multi-field Hospital,Kharkiv, Ukraine). Participants were not compensated to participate in this trial.
Period: Overall Study
Arm/Group | L-Alanyl/L-Glutamine- Laparoscopic | Physiological Saline- Laparoscopic | L-Alanyl/L-Glutamine- Laparotomy | Physiological Saline- Laparotomy
Started | 18 | 19 | 5 | 5
Completed | 15 | 17 | 4 | 3
Not Completed | 3 | 2 | 1 | 2
Not completed — Withdrawal by Subject | 2 | 2 | 1 | 2
Not completed — Adverse Event | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | L-Alanyl/L-Glutamine- Laparoscopic | Physiological Saline- Laparoscopic | L-Alanyl/L-Glutamine- Laparotomy | Physiological Saline- Laparotomy | Total
Number analyzed (Participants) | 18 | 19 | 5 | 5 | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 18 | 19 | 5 | 5 | 47
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 19 | 5 | 5 | 47
  Male | 0 | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 23.5 (4.3) | 22.3 (3.0) | 24.5 (7.9) | 23.5 (3.5) | 23.5 (0.9)
Temperature (Degrees Celsius) [Mean (Standard Deviation); unit: Degrees Celsius] | 36.7 (0.1) | 36.3 (0.1) | 36.7 (0.1) | 36.6 (0.1) | 36.5 (0.2)
Heart rate (bpm) [Mean (Standard Deviation); unit: beats per minute] | 79.8 (8.6) | 79.4 (7.6) | 79 (1.8) | 73 (8.3) | 77.8 (3.2)
Systolic BP (mmHg) [Mean (Standard Deviation); unit: mmHg] | 113.9 (9.5) | 113.9 (8.6) | 117 (5.7) | 110 (10) | 113.7 (2.9)
Diastolic BP (mmHg) [Mean (Standard Deviation); unit: mmHg] | 70.0 (5.0) | 70.3 (6.1) | 71 (2.2) | 67 (6.7) | 69.6 (1.8)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants in Which Adhesions Were Prevented.
Description: The American Fertility Society (AFS) grading system for adhesions was used to assess incidence of adhesions. Adhesion prevention was determined through grading of adhesions at the time of myomectomy (initial surgery) and at the time of second look surgery and compared.
Time Frame: 6-8 weeks
Population: The number of subjects in each study group (Control [N=20] and AG [N=19]) was lower at the second look laparoscopic (SLL) compared to the number of subjects originally enrolled in each study group. The difference between groups numbers is a result of dropouts, including subjects who failed criteria for SLL or who elected not to continue the study. The laparotomy group, given the small sample size, was primary used to gather safety data.
Measure: Count of Participants; unit: Participants
Arm/Group | L-Alanyl/L-Glutamine- Laparoscopic | Physiological Saline- Laparoscopic | L-Alanyl/L-Glutamine- Laparotomy | Physiological Saline- Laparotomy
Number analyzed (Participants) | 15 | 17 | 4 | 3
Participants | 15 | 5 | 4 | 3

2. Secondary Outcome: Adverse Events, Adverse Drug Reactions and Clinical Laboratory Abnormalities.
Description: Participants With Treatment-related Adverse Events as Assessed by Clinical Blood Work Abnormalities and Physical Examination.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Groups:
- L-Alanyl/L-Glutamine: Participants receiving intraperitoneal administration of L-Alanyl-L-Glutamine at the time of laparoscopic myomectomy.
  L-Alanyl/L-Glutamine: Sterile solution of L-Alanyl-L-Glutamine, 400mg/mL in water for injection. It is dosed at 1g/kg of body weight and is instilled into the peritoneum at the time of surgery. The active ingredient, glutamine, is a conditionally essential amino acid component of nutritional supplements.
- Physiological Saline: Participants receiving intraperitoneal administration of physiological saline at the time of laparoscopic myomectomy.
  Physiologic saline: Placebo
Arm/Group | L-Alanyl/L-Glutamine | Physiological Saline | L-Alanyl/L-Glutamine- Laparotomy | Physiological Saline- Laparotomy
Number analyzed (Participants) | 18 | 19 | 5 | 5
Participants | 3 | 6 | 1 | 1

ADVERSE EVENTS:
Time Frame: Adverse events were monitored for 8 weeks post-myomectomy.
Description: Safety was assessed though the incidence of adverse drug events (AE) and clinical lab abnormalities. The laparotomy arms were included for safety analysis, and laboratory assessments were conducted at the time of myomectomy and at SLL for all patients that enrolled and completed the study.
Groups:
- Physiological Saline -Laparotomy: Participants receiving intraperitoneal administration of physiological saline at the time of myomectomy (laparotomy).
  Physiologic saline: Placebo
Arm/Group | L-Alanyl/L-Glutamine- Laparoscopic | Physiological Saline- Laparoscopic | L-Alanyl/L-Glutamine- Laparotomy | Physiological Saline -Laparotomy
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/19 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/19 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 3/18 | 6/19 | 1/5 | 1/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | L-Alanyl/L-Glutamine- Laparoscopic (N=18) | Physiological Saline- Laparoscopic (N=19) | L-Alanyl/L-Glutamine- Laparotomy (N=5) | Physiological Saline -Laparotomy (N=5)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Elevated AST levels (Hepatobiliary disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) — aspartate aminotransferase (AST)
Elevated temperature (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Elevated CPK levels (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) — creatine phosphokinase (CPK)

LIMITATIONS AND CAVEATS:
There were no limitations and caveats to the trial that would impact the integrity, analysis or interpretation of the trial results. Dropouts were accounted for in the study design and those excluded did not impact the statistics and/or the power of the trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No